CLINICAL TRIAL: NCT01446887
Title: Phase II Study of Prophylactic Anticoagulation for Preventing Deep Vein Thrombosis After Total Hip Arthroplasty
Brief Title: Prophylactic Anticoagulation for Preventing Deep Vein Thrombosis After Total Hip Arthroplasty
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: JIANG Qing (Other)
Responsible Party: Sponsor-Investigator, JIANG Qing, Director, The Center of Diagnosis and Treatment for Joint Disease, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Organization: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NJDVTS
Record Dates: First submitted 2011-09-28; First posted 2011-10-05 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Deep Vein Thrombosis
Keywords: Deep Vein Thrombosis; total hip arthroplasty; prophylactic anticoagulation; randomized study
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- non-prophylactic anticoagulation (No Intervention): without prophylactic anticoagulation
- prophylactic anticoagulation (Experimental): prophylactic anticoagulation by rivaroxaban
  Interventions: Other: prophylactic anticoagulation

INTERVENTIONS:
Other: prophylactic anticoagulation — prophylactic anticoagulation by rivaroxaban
  Arms: prophylactic anticoagulation

SUMMARY:
Deep vein thrombosis (DVT) remains a life-threatening complication of arthroplasty. It remains controversial for anticoagulation strategies after total hip arthroplasty (THA). A randomized double-blind study was conducted to determine whether prophylactic anticoagulation was efficient reduce DVT after THA. subjects who underwent uncemented THA were assigned to prophylactic anticoagulation group or non- prophylactic anticoagulation group. Patients were followed up 3 months later after surgery. DVT was tested by contrast venography. Investigator also used logistic regression analysis with variable selection for obtaining the prediction model of DVT. DVT after THA was affected by personal (age) and clinical factors (mechanical compression, duration of surgery). THA with short duration of surgery did not require prophylactic anticoagulation.

ELIGIBILITY:
Inclusion Criteria:

* Primary total hip arthroplasty

Exclusion Criteria:

* Revision hip replacement, total knee replacement, revision knee replacement, semi-hip replacement and cemented THR were excluded.
* Coagulation related disease and cancer were excluded either.

Ages: 35 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-01; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
all cause DVT | 7 days
  deep-vein thrombosis nonfatal pulmonary embolism, or death

SECONDARY OUTCOMES:
Major DVT | 7 days
  major venous thromboembolism (proximal deep-vein thrombosis, nonfatal pulmonary embolism, or death from venous thromboembolism)

CONTACTS AND LOCATIONS:
Locations (1):
- The Center of Diagnosis and Treatment for Joint Disease, Drum Tower Hospital, Nanjing, Jiangsu, China